CLINICAL TRIAL: NCT00001093
Title: Outcomes of Antiretroviral Therapy During Primary HIV Infection
Brief Title: Outcomes of Anti-HIV Therapy During Early HIV Infection
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Other Study IDs: AI-05-005; AEHIV 005; AIEDRP AI-05-005
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: HIV Infections
Keywords: Immunity, Cellular; Sexual Partners; Treatment Outcome; Anti-HIV Agents; Viral Load; Acute Infection
MeSH Terms: conditions — HIV Infections

SUMMARY:
The purpose of this study is to find out if it is effective to give aggressive anti-HIV therapy to patients who have been infected recently with HIV.

Many doctors recommend that patients who have recently been infected with HIV begin anti-HIV treatment as soon as possible. However, early HIV infection is not yet completely understood, so it is not known if this is the best approach. This study will look at the effects of beginning anti-HIV treatment during early HIV infection.

DETAILED DESCRIPTION:
Although many researchers have recommended initiation of aggressive antiretroviral therapy as soon as possible after HIV infection occurs, the tolerability and efficacy of this approach has not been systemically evaluated. Many features of primary HIV pathogenesis are incompletely understood. A more complete understanding of immune dynamics and viral pathogenesis during primary HIV infection is critical to determine optimal treatment intervention strategies. This study will evaluate the outcomes of potent antiretroviral therapy initiated at different stages of primary HIV infection.

Thirty-six of the study patients are coenrolled to ACTG 371 or another treatment protocol. All study drug treatment and toxicity management is performed according to guidelines in these treatment protocols. An untreated cohort of 12 patients is also followed on this study. Patients are stratified at enrollment according to their stage of acute or early HIV infection. Patients are evaluated for virologic, immunologic, and clinical parameters for 96 weeks. In addition, novel studies of source partner identification are proposed. An effort is made to determine the most likely source partner(s) for each study patient on the basis of patient recall of possible exposures. A separate study protocol will evaluate the source partner.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are at least 13 years old.
* Have acute or early HIV infection. The stage of HIV infection will depend on the results from certain lab tests.

Exclusion Criteria

Patients will not be eligible for this study if they:

* Are pregnant or breast-feeding.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48
Dates: Start 1999-10; Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Little, Principal Investigator; James Kahn, Principal Investigator; Eric Daar, Principal Investigator
Locations (3):
- United States (3):
  - Cedars Sinai Med Ctr, Los Angeles, California
  - UCSD, San Diego, California
  - San Francisco Gen Hosp / UCSF AIDS Program, San Francisco, California